CLINICAL TRIAL: NCT01558089
Title: Ability To Achieve A Good Eular Response In Patients With Moderate-to-severe Active Early Rheumatoid Arthritis Who Satisfy The New Acr/Eular Classification Criteria Receiving Etanercept + Mtx In Real World Clinical Practice In Greece
Brief Title: Good EULAR Response In Patients With Early Rheumatoid Arthritis
Acronym: EARLY RA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801138
Record Dates: First submitted 2012-02-15; First posted 2012-03-20 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- etanercept + methotrexate
  Interventions: Drug: etanercept; Drug: methotrexate

INTERVENTIONS:
Drug: etanercept — according to SmPC and clinical practice
Drug: methotrexate — according to SmPC and clinical practice

SUMMARY:
This open-label, prospective, observational study will evaluate the clinical response to etanercept + methotrexate therapy in patients with moderate to severe rheumatoid arthritis, as prescribed by the rheumatologist in a normal clinical setting in Greece

DETAILED DESCRIPTION:
All subjects enrolled should meet the usual prescribing criteria for Etanercept as per the local product information and should be entered into the study at the investigator's discretion

ELIGIBILITY:
Inclusion Criteria:

1. signed and dated informed consent document
2. 18 years of age and older at the time of consent
3. Patients with moderate-to-severe active rheumatoid arthritis, who satisfy the 2010 Rheumatoid Arthritis Classification Criteria
4. Patients who have been prescribed for first time to receive treatment with MTX + Etanercept prior to enrollment to this study, following routine clinical practice and according to the approved SmPC,
5. Patients with DAS28 ≥ 3.2
6. Duration of disease symptoms ≥ 6 weeks and ≤2 years
7. Failure to respond to prior DMARDs including MTX monotherapy according to routine clinical practice.

Exclusion Criteria:

1. Contraindications according to the SmPC
2. History of or present anti-TNFa or other biologic therapy for the treatment of RA
3. Known significant concurrent medical disease according to investigator's opinion and the current SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with rheumatoid arthritis who fulfill the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2013-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Greece (9):
  - G. Gennimatas General Hospital /Rheumatology Clinic, Athens, Attica
  - Ippokrateio General Hospital of Athens / 2nd internal Medicine Clinic of the University of Athens, Athens, Attica
  - University General Hospital of Heraklion, Heraklion, Creete
  - G. Papanikolaoy, Thessaloniki, Exochi
  - 424 Military Hospital, Thessaloniki, Thessalonikis
  - Euromedica Kyanous Stavros, Thessaloniki, Thessaloniki
  - Laiko General Peripheral Hospital, Athens
  - Peripheral University General Hospital of Larissa, Larissa
  - "Olympion therapeutic center" General Clinic of Patras, Pátrai

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801138&StudyName=Good%20EULAR%20response%20in%20patients%20with%20early%20rheumatoid%20artrhitis

RESULTS

PARTICIPANT FLOW:
Groups:
- ETANERCEPT/ METHOTREXATE: The study group comprised adult patients who at the time of entry had moderate-to-severe rheumatoid arthritis (RΑ), having symptoms for at least 6 weeks and no more than 2 years while satisfying the 2010 RA classification criteria, Disease Activity Score 28 (DAS28) ≥3.2, and who were prescribed for the first time to receive Methotrexate + Etanercept according to routine clinical practice and current summary of product characteristics, prior to enrollment in this study.
Period: Overall Study
Arm/Group | ETANERCEPT/ METHOTREXATE
Started | 76
Completed | 63
Not Completed | 13
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | ETANERCEPT/ METHOTREXATE
Number analyzed (Participants) | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Primary: Participants With EULAR (Good)
Description: Good European League Against Rheumatism (EULAR) response at 6 months based on DAS28 EULAR response criteria defined as Good response = DAS28 change >1.2 with DAS28 ≤3.2; Moderate response = DAS28 change >0.6 with DAS28 >3.2-5.1; Non-response = DAS28 change ≤0.6 and absolute DAS28 >5.1
Time Frame: Visit 4 (Month 6)
Population: Last observation carried forward (LOCF) was applied where data were available. Participants where a EULAR response value could not be calculated, were omitted from the analysis. Only 48 Participants had available EULAR response data at 6 months.
Measure: Number; unit: participants
Groups:
- Etanercept/Methotrexate: All participants in this study who received Etanercept and Methotrexate
Arm/Group | Etanercept/Methotrexate
Number analyzed (Participants) | 48
participants | 19

2. Secondary Outcome: Change From Baseline in Tender Joint Count at Visit 4 (Month 6)
Description: In order to calculate the DAS28 the number of swollen joints and tender joints were assessed using the 28 Joint Count (TJC28 and SJC28). A joint was counted as tender/swollen if the tender/swelling code was 'Present'. Swollen and tender 28 joint counts will be performed at visit 1 (baseline), visit 2, visit 3 and visit 4 or early withdrawal.
Time Frame: Baseline and Visit 4 (Month 6)
Population: The analysis was based on the Full Analysis Set (FAS) population. The FAS comprised participants who received at least 1 dose of Methotrexate + Etanercept, and completed at least 1 assessment following first dose.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept/Methotrexate
Number analyzed (Participants) | 63
Joints | -7.68 (7.08)

3. Secondary Outcome: Change From Baseline in Swollen Joint Count at Visit 4 (Month 6)
Description: as for outcome 2
Time Frame: Baseline and Visit 4 (Month 6)
Population: The analysis was based on the FAS population. The FAS comprised participants who received at least 1 dose of Methotrexate + Etanercept, and completed at least 1 assessment following first dose.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Etanercept/Methotrexate
Number analyzed (Participants) | 63
Joints | -4.52 (5.22)

4. Secondary Outcome: Change From Baseline in Patient's Assessment of General Health (VAS) at Visit 4 (Month 6)
Description: The patients used a 100 mm Visual Analogue Scale (VAS) to score their general health during the last week. The scale ranged from 0 (no pain) to 100 mm (severe pain)
Time Frame: Baseline and Visit 4 (Month 6)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Etanercept/Methotrexate
Number analyzed (Participants) | 44
mm | -38.14 (28.79)

5. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Visit 4 (Month 6)
Time Frame: Baseline and Visit 4 (Month 6)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Etanercept/Methotrexate
Number analyzed (Participants) | 38
mm/hour | -21.21 (22.28)

6. Secondary Outcome: Change From Baseline in EQ-5D Health Index at Visit 4 (Month 6)
Description: The European Quality of Life-5 Dimensions (EQ-5D) was measured on a 5 item scale. The scores for the 5 items (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) ranged from 1 (no problem) to 3 (extreme problems). For EQ-5D, participants rate questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. Each of the 5 dimensions is divided into 3 levels of perceived problems: Level 1=no problem; level 2=some problem; level 3=extreme problem. A unique health state is defined by combining 1 level from each dimension. A total of 243 possible health states are defined in this way. Each state is referred to in terms of a 5 digit code. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline and Visit 4 (Month 6)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept/Methotrexate
Number analyzed (Participants) | 49
units on scale | 0.40 (0.36)

7. Secondary Outcome: Change From Baseline in HAQ-DI at Visit 4 (Month 6)
Description: The Health Assessment Questionnaire-Disability Index (HAQ-DI) is composed of 20 items. It is a participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; common activities over past week. Each item scored on 4-point scale from 0-3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as sum of domain scores and divided by number of domains answered. Total possible score ranges from 0-3: 0=least difficulty and 3=extreme difficulty.
Time Frame: Baseline and Visit 4 (Month 6)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Etanercept/Methotrexate
Number analyzed (Participants) | 52
units on scale | -0.78 (0.63)

8. Secondary Outcome: Predictor of Good EULAR Response Versus Moderate/No Response at Visit 4 (Month 6) - DAS28 (LOCF)
Description: In a first step a univariate logistic regression model was fit for the following baseline variables: DAS28 (n=48), Physician's Global Assessment of Disease Activity (VAS) (n=47), Patient's Global Assessment of Disease Activity (VAS) (n=47), CRP (n=46), Patient Pain (VAS) (n=47), HAQ-DI (n=47), EQ-5D (n=47). Only those variables that were significant at a 10% level were then included in the second step: a multivariate analysis with stepwise regression (entry level=10%, stay level=5%). The final model presented in the Basic Results table displays those covariates which were significant at the 2-sided 5% level (baseline value for DAS28; n=48). Note that DAS28 is not a categorical variable; therefore no stratified results for this variable are presented.
Time Frame: Baseline and Visit 4 (Month 6)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Odds Ratio (per unit increase)
Arm/Group | Etanercept/Methotrexate
Number analyzed (Participants) | 48
Odds Ratio (per unit increase) | 2.831 [1.358 to 5.898]

ADVERSE EVENTS:
Arm/Group | ETANERCEPT/ METHOTREXATE
Serious Adverse Events (participants affected / at risk) | 6/76
Other Adverse Events (participants affected / at risk) | 14/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETANERCEPT/ METHOTREXATE (N=76)
Ulcerative keratitis (Eye disorders) | 1
Injection site pruritus (General disorders) | 1
Gallbladder disorder (Hepatobiliary disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ETANERCEPT/ METHOTREXATE (N=76)
Vertigo (Ear and labyrinth disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Drug ineffective (General disorders) | 2
Injection site erythema (General disorders) | 2
Injection site pruritus (General disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.